CLINICAL TRIAL: NCT06969599
Title: The Impact of Bedtime Screen Use on Sleep Quality and Cognitive Function in Medical Graduate Students: A Cross Sectional Correlation Study
Brief Title: A Cross-sectional Study on the Correlation Between Screen Usage and Sleep and Cognition in Medical Students
Status: Not yet recruiting | Type: Observational
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: NFEC-2025-144
Record Dates: First submitted 2025-04-28; First posted 2025-05-14 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Sleep Quality
Keywords: sleep
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — stool specimen
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: No intervention measures — No intervention measures

SUMMARY:
The aim of this study is to investigate the effects of screen use within one hour before bedtime on sleep quality and cognitive function in medical graduate students, and to verify the mediating effect of sleep quality between the two. The study adopted a cross-sectional observational design and planned to enroll 508 full-time medical graduate students. The primary endpoints were evaluated using the Pittsburgh Sleep Quality Index (PSQI) and standardized cognitive tests (N-back, ANT, etc.), while secondary endpoints included insomnia severity, anxiety/depression regulation, gut microbiota diversity, and the interaction between physical activity and sleep. Data collection includes questionnaire surveys (PSQI, ISI, GAD-7, etc.), cognitive task testing, and analysis of gut microbiota samples. The final result will provide scientific basis for improving the sleep and cognitive health of medical graduate students.

ELIGIBILITY:
1. Inclusion criteria:

   1. Full time medical graduate student at Southern Medical University
   2. Age ≥ 18 years old
2. Exclusion criteria:

   1. Have taken the following medications within the past month: antibiotics, probiotics, sleeping pills, laxatives, or intestinal cleansers, etc;
   2. Serious gastrointestinal diseases (inflammatory bowel disease, Crohn's disease, gastric cancer, etc.);
   3. Recently (within one month) experienced major life events (such as the death of a relative, surgery);

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: medical postgraduate
Sampling Method: Non-Probability Sample
Enrollment: 508 (Estimated)
Dates: Start 2025-05-15 (Estimated); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
Sleep questionnaire cognitive task | baseline
  Sleep quality assessed through the Pittsburgh Sleep Quality Index (PSQI) total score,The higher the PSQI score, the more likely it is that the sleep quality is poor

IPD SHARING:
Plan to Share IPD: Yes
论文
Supporting Information: Study Protocol, SAP